CLINICAL TRIAL: NCT07113366
Title: Improvement of Atopic Dermatitis Symptoms and Signs by Jelly Fig (Ficus Awkeotsang Makino) Extract
Brief Title: Efficacy of Jelly Fig (Ficus Awkeotsang Makino) Extract for Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chiau-Sheng Jang, Department of Dermatology, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan., Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSVGH24-CT3-31
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose FAE cream (5.0 mg/mL) (Active Comparator): Ficus awkeotsang Makino extract (FAE)
  Interventions: Drug: FAE cream
- Low- dose FAE cream (1.0 mg/mL) (Active Comparator): Ficus awkeotsang Makino extract (FAE)
  Interventions: Drug: FAE cream
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FAE cream — Ficus awkeotsang Makino extract (FAE)
  Arms: High-dose FAE cream (5.0 mg/mL); Low- dose FAE cream (1.0 mg/mL)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the efficacy and safety of a topical formulation containing Ficus awkeotsang Makino extract (FAE), derived from jelly fig, in participants with mild to moderate atopic dermatitis. Ficus awkeotsang is a traditional plant native to Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years at the time of enrollment
* Clinical diagnosis of atopic dermatitis (AD) according to the Hanifin and Rajka criteria
* Investigator's Global Assessment (IGA) score of 2 (mild) or 3 (moderate) at screening

Exclusion Criteria:

* Prior treatment with biologic agents within 16 weeks before baseline
* Use of phototherapy, systemic corticosteroids, or other systemic immunosuppressants within 28 days before baseline
* Use of topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 14 days before baseline
* Presence of active skin infections
* Pregnancy or breastfeeding
* Known hypersensitivity to any component of the investigational product

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Investigator's Global Assessment (IGA) Success | Day 28
  IGA success is defined as achieving a score of 0 (clear) or 1 (almost clear) with a ≥2-point improvement from baseline on the 5-point IGA scale. The scale ranges from 0 (clear) to 4 (severe), with lower scores indicating less disease severity.
  Unit of Measure: Percentage of participants (%)

SECONDARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) Score from Baseline to Days 7 and 28 | Baseline, Day 7, and Day 28
  The EASI score ranges from 0 to 72, with higher scores indicating more severe disease. This outcome measures the change in EASI score from baseline.
  Unit of Measure: Units on a scale
Change in Peak Pruritus Numerical Rating Scale (pp-NRS) Score from Baseline to Days 7 and 28 | Baseline, Day 7, and Day 28
  The pp-NRS is an 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Participants rate their worst itch over the past 24 hours.
  Unit of Measure: Units on a scale
Change in Body Surface Area (BSA) Affected by Atopic Dermatitis from Baseline to Days 7 and 28 | Baseline, Day 7, and Day 28
  This outcome measures the percentage of body surface area affected by atopic dermatitis.
  Unit of Measure: Percent (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided